CLINICAL TRIAL: NCT05494437
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Multiple-Dose, Placebo Controlled Clinical Trial of Two Doses of PP-01 for the Mitigation of Cannabis Withdrawal Symptoms
Brief Title: Effect of PP-01 on Cannabis Withdrawal Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PleoPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAN-002
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Cannabis Withdrawal
Keywords: Cannabis Use Disorder; Marijuana Use Disorder
MeSH Terms: interventions — nabilone; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- PP-01 High Dose (Experimental): Oral PP-01 High Dose tapered/titrated over 34 days
  Interventions: Combination Product: PP-01 High Dose
- PP-01 Low Dose (Experimental): Oral PP-01 Low Dose tapered/titrated over 34 days
  Interventions: Combination Product: PP-01 Low Dose
- Placebo (Placebo Comparator): Oral placebo, given daily for 34 days
  Interventions: Drug: Placebo
- Nabilone (Active Comparator): oral nabilone, tapered/titrated over 28 days
  Interventions: Drug: Nabilone
- Gabapentin (Active Comparator): oral gabapentin, tapered/titrated over 34 days
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Combination Product: PP-01 High Dose — Cannabinoid-1 (CB1) partial agonist / GABAergic modulator
  Arms: PP-01 High Dose
Combination Product: PP-01 Low Dose — CB1 partial agonist / GABAergic modulator
  Arms: PP-01 Low Dose
Drug: Placebo — Placebo comparator
  Arms: Placebo
Drug: Nabilone — CB1 receptor
  Arms: Nabilone
Drug: Gabapentin — GABAergic modulator
  Arms: Gabapentin

SUMMARY:
This study will be a randomized, double-blind, placebo-controlled, multicenter trial conducted to evaluate whether PP-01 mitigates the withdrawal symptoms associated with discontinuing cannabis in participants with moderate to severe Cannabis Use Disorder (CUD). The study will enroll approximately 225 participants with moderate to severe CUD and will include 5 arms, including a placebo arm, to help assess the incidence and severity of withdrawal symptoms in heavy long-term users of cannabis. Participants receive study medication for 34 days and participate in 11 visits (7 at a clinic and 4 telemedicine).

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy individuals between the ages of 18 and 55, inclusive
2. Meets Diagnostic and Statistical Manual (DSM)-5 diagnostic criteria for current moderate to severe CUD as confirmed by a licensed physician or psychologist or addiction medicine specialist
3. BMI within 18.0 to 38.0 kg/m2, inclusive
4. Seeking to minimize withdrawal symptoms related to cannabis discontinuation in people seeking to discontinue cannabis
5. Meet DSM-5 Cannabis Withdrawal
6. Report heavy use of daily/near daily cannabis
7. Have a urine drug screen positive for tetrahydrocannabinol (THC)/THC metabolites at Screening and Randomization
8. Capable of giving informed consent and complying with study procedures
9. Stated willingness to comply with all study procedures including twice weekly visits, daily evening video calls, restrictions, and availability for the duration of the study

Exclusion Criteria:

1. Lifetime history of DSM-5 diagnosis of schizophrenia or schizoaffective disorder, or Bipolar 1 within the previous 2 years
2. Current DSM-5 criteria for a psychiatric disorder that in the Investigator's judgment is unstable, would be disrupted by the study medication, or is likely to require new pharmacotherapy or psychotherapy during the study period. Individuals who are currently stable on psychotropic medication for at least 3 months may be included at the discretion of the Investigator's judgement
3. Participants who meet DSM-5 criteria for any substance use disorder other than cannabis, nicotine, or caffeine use disorders
4. Participants using cannabis for a medical condition requiring use such as epilepsy
5. Clinically significant unstable medical disorders
6. Any clinically important abnormalities on Screening physical examination (PE), assessments, ECG, or laboratory tests
7. Use of an investigational drug or biologic within 30 days or 5 times the half-life (whichever is longer) prior to the Screening Visit
8. Pregnant or lactating female participants, or a positive urine pregnancy test
9. COVID-19

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of a patient reported outcome measure of cannabis withdrawal over 5 days | Over 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Jay Constantine, MD, Study Director — PleoPharma, Inc.
Locations (18):
- United States (18):
  - Behavioral Research Specialists, LLC, Glendale, California
  - Synergy San Diego, Lemon Grove, California
  - Neuropsychiatric Research Institute, Orange, California
  - CNS Clinical Research Group, Coral Springs, Florida
  - Gulf Coast Clinical Research, Fort Myers, Florida
  - Innovative Clinical Research Inc., Lauderhill, Florida
  - CenExel iResearch Atlanta, LLC, Decatur, Georgia
  - CenExel iResearch Savannah, LLC, Savannah, Georgia
  - Pillar Clinical Research, LLC, Chicago, Illinois
  - Otrimed Research Center, Edgewood, Kentucky
  - Tandem Clinical Research, Marrero, Louisiana
  - Benchmark Research, Shreveport, Louisiana
  - Hassman Research Institute, Berlin, New Jersey
  - North Star Medical Research, Middleburg Heights, Ohio
  - Pahl Pharmaceutical Professionals LLC, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Austin Clinical Trials, Austin, Texas
  - Cedar Clinical Research, Draper, Utah

IPD SHARING:
Plan to Share IPD: No